CLINICAL TRIAL: NCT04993846
Title: Pancreatic canceR pErioDontAl sTatus and Oral micRobiome - PREDATOR Study
Brief Title: Pancreatic Cancer and Oral Microbiome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: 3292CESC
Record Dates: First submitted 2021-05-26; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-01

CONDITIONS: Oral Microbiome; Pancreatic Cancer; IPMN; Parodontopathy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Pancreatic cancer patients - Explorative phase: Pancreatic cancer patients evaluated at the Pancreatic Surgery Unit of the Pancreas Institute of the University of Verona will be enrolled. Fifteen PC patients per stage will be selected (15 Stage I/II, Stage III, Stage IV). Patients may have been scheduled for surgery or for biopsy for future systemic treatments. An oral microbiota (dental plaque) sample will be collected and a periodontal and dental assessment will be performed, before any therapeutic procedure, together with orthopantomography
  Interventions: Diagnostic Test: Dental plaque sampling; Diagnostic Test: qPCR
- Healthy controls - Explorative phase: Age-matched (+- 5 years) healthy controls referring to the Odontostomatology Unit for oral procedure according to clinical practice, with a recent (not longer than 12 months) cross-sectional abdominal imaging excluding gastrointestinal cancers.
  Interventions: Diagnostic Test: Dental plaque sampling; Diagnostic Test: qPCR
- Pancreatic cancer patients - Validation phase: Pancreatic cancer patients evaluated at the Pancreatic Surgery Unit of the Pancreas Institute of the University of Verona will be enrolled. Fifteen PC patients per stage will be selected (15 Stage I/II, Stage III, Stage IV). Patients may have been scheduled for surgery or for biopsy for future systemic treatments.
  Interventions: Diagnostic Test: Dental plaque sampling; Diagnostic Test: qPCR
- Healthy controls - Validation phase: Age-matched (+- 5 years) healthy controls referring to the Odontostomatology Unit for oral procedure according to clinical practice, with a recent (not longer than 12 months) cross-sectional abdominal imaging excluding gastrointestinal cancers.
  Interventions: Diagnostic Test: Dental plaque sampling; Diagnostic Test: qPCR
- IPMN patients controls - Validation phase: Patients suffering from IPMNs evaluated at outpatients clinics or scheduled for surgery.
  Interventions: Diagnostic Test: Dental plaque sampling; Diagnostic Test: qPCR

INTERVENTIONS:
Diagnostic Test: Dental plaque sampling — Dental plaque sampling
Diagnostic Test: qPCR — qPCR

SUMMARY:
Pancreatic cancer (PC) is a solid malignancy with a dismal prognosis. It has a 5-year survival rate of approximately 8%. This is due to the usually late diagnosis, to chemoresistance, and to intrinsic biological aggressiveness. Risk factors for PC are smoking, alcohol, chronic pancreatitis, obesity, and diabetes. Recently, research has been dedicated to the identification of a causal connection between certain pathogenic microorganisms, especially of the oral flora, and PC. This would ultimately allow to identify new biomarkers to adopt for early diagnosis, or to create new strategies for prevention.

Oral microbiota, periodontal disease and neoplastic risk

When referring to "oral microbiota" (OM), about 700 hundreds bacterial species are mentioned, colonizing the oral cavity. A change in the normal flora of the oral cavity is commonly indicated with the term "dysbiosis".

The causal connection between oral microbiota, periodontal disease and neoplastic risk is possibly triple. First, it has been found that oral flora substantially differentiates between cancer patients and controls. In particular, the most predominant phyla in cancer patients are Firmicutes and Actinobacteria, whereas Proteobacteria, Fusobacteria, and Bacteroides are more common in healthy controls. This highlights the possibility of a direct causal connection between dysbiosis and neoplastic risk. Second, oral dysbiosis represents the main risk factor of PD that per sé is a risk factor of many cancers. Third, the conditions leading to oral dysbiosis (alcohol, smoking, obesity, diabetes, chronic drugs intake, dietary habits, etc.) are the most well known risk factors either for cancer and oral dysbiosis. The common denominator is always represented by chronic inflammation and migration of microorganisms to distant sites, ultimately promoting neoplastic progression.

This tangled net of causal connections sheds light on the potential important role of the oral cavity and PD as independent risk factors for many cancers, and as modifiable elements to reduce the neoplastic risk and to perform prevention(15).

Oral microbiota, periodontal disease and pancreatic cancer

In 2012, the pioneering study by Farrell et al. showed that bacteria of the OM can discriminate PC patients from healthy subjects. Since then, few other studies have shown that changes of the OM are independent risk factors for PC and that the OM of PC patients differs than controls. The involved bacterial species are many and their role seems to be contrasting on the basis of the study considered. Farrell et al. found that the combined adoption of Neisseria elongata and Streptococcus mitis distinguished PC patients from healthy controls (both showed low levels in PC patients, AUC of combined sensitivity 0.9), and that higher levels of Granulicatella adiacens and Streptococcus Mitis distinguished PC patients from chronic pancreatitis ones. Torres et al. found a higher ratio of Leptotrichia to Porphyromonas in PC patients. Fan et al. reported that Porphyromonas gingivalis, Prevotella intermedia, Alloprevotella and Aggregatibacter actinomycetemcomitans are associated with a higher risk of PC, whereas Fusobacteria and Leptotrichia were associated with a decreased risk. Another study evaluating the diversity of OM in three groups of individuals (PC patients, patients suffering from Intraductal papillary mucinous neoplasms [a pancreatic preneoplastic condition], and healthy controls), excluding current smokers and users of antibiotics, found no differences in the OM, although patients with PC had a higher proportion of Firmicutes compared with Intraductal Papillary Mucinous Neoplasms (IPMNs) and controls. Lastly, a recent study by Gaiser et al. showed that the cystic fluid of patients submitted to surgery for IPMNs contained bacterial species that are commonly found in the oral cavity, including, among the others, Granulicatella adiacens, Fusobacterium nucleatum. These two, in particular, were higher in the cohort of individuals with IPMNs with high-grade dysplasia, indicating a pivotal role in tumorigenesis(19).

As regards PD, the first studies demonstrating an association between PD and PC date back to the mid of 2000's, and they were confirmed afterward, even adjusting confounders such as diabetes, pancreatitis, hyperlipemia, smoking or alcohol-related conditions. PD is strictly connected to oral hygiene, that seems to be associated to an increased risk of PC. It is now clear that PD can concur to development of PC in several ways, promoting chronic inflammation, spreading continuously to distant organs (including pancreas) pro-tumorigenic bacteria, or promoting a chronic alteration of the immune function that make the individual more prone to develop a cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years;
* The ability of the subject to understand the character and individual consequences of the clinical trial
* Written informed consent

Exclusion Criteria:

* A recent history of antibiotics (< 4 weeks before the enrolment)
* Current systemic or topic medication with steroids
* Active smoking or alcohol habits
* Vegan diet or dietary disorders (anorexia, bulimia)
* Immune system disorders
* Diabetes
* Obesity (defined as having a BMI > 30)
* Other current malignancies
* History of gastrointestinal tract resections, chronic gastrointestinal diseases (es. Inflammatory bowel diseases, or gastroesophageal reflux disease)
* Pregnant or breastfeeding patients
* Impaired mental state or language problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a cyto-histological diagnosis of pancreatic cancer, respecting the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative analysis of the dental plaque microbiome in patients with pancreatic cancer vs. healthy controls and IPMN patients | Baseline (At enrollment)
  Whole-Genome Sequencing analysis
Correlation analysis between periodontal status and dental plaque microbiome | Baseline (At enrollment)
  According to the periodontal status (appropriate scores will be used), patients will be divided into distinct groups. The proportional means of abundance of selected genera and species, and bacterial load (real-time data) between these groups will be analyzed using the Mann-Whitney U-test. Correlations between mean distributions of the genera and species and the parodontal status scores values will be analysed using the Spearman Correlation Coefficient.
Quantitative analysis of the dental plaque microbiome in patients with pancreatic cancer vs. healthy controls and IPMN patients | Baseline (At enrollment)
  Whole-Genome Sequencing analysis

SECONDARY OUTCOMES:
Qualitative analysis of OM and periodontal status between the various stages of PC | Baseline (At enrollment)
  Whole-Genome Sequencing analysis

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - General and Pancreatic Surgery Unit, Verona
  - Section of Dentistry and Maxillofacial Surgery, Department of Surgical Sciences, Paediatrics and Gynaecology, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fan X, Alekseyenko AV, Wu J, Peters BA, Jacobs EJ, Gapstur SM, Purdue MP, Abnet CC, Stolzenberg-Solomon R, Miller G, Ravel J, Hayes RB, Ahn J. Human oral microbiome and prospective risk for pancreatic cancer: a population-based nested case-control study. Gut. 2018 Jan;67(1):120-127. doi: 10.1136/gutjnl-2016-312580. Epub 2016 Oct 14. PMID 27742762
- [Result] Farrell JJ, Zhang L, Zhou H, Chia D, Elashoff D, Akin D, Paster BJ, Joshipura K, Wong DT. Variations of oral microbiota are associated with pancreatic diseases including pancreatic cancer. Gut. 2012 Apr;61(4):582-8. doi: 10.1136/gutjnl-2011-300784. Epub 2011 Oct 12. PMID 21994333
- [Result] Torres PJ, Fletcher EM, Gibbons SM, Bouvet M, Doran KS, Kelley ST. Characterization of the salivary microbiome in patients with pancreatic cancer. PeerJ. 2015 Nov 5;3:e1373. doi: 10.7717/peerj.1373. eCollection 2015. PMID 26587342
- [Result] Olson SH, Satagopan J, Xu Y, Ling L, Leong S, Orlow I, Saldia A, Li P, Nunes P, Madonia V, Allen PJ, O'Reilly E, Pamer E, Kurtz RC. The oral microbiota in patients with pancreatic cancer, patients with IPMNs, and controls: a pilot study. Cancer Causes Control. 2017 Sep;28(9):959-969. doi: 10.1007/s10552-017-0933-8. Epub 2017 Jul 31. PMID 28762074
- [Result] Michaud DS, Izard J, Wilhelm-Benartzi CS, You DH, Grote VA, Tjonneland A, Dahm CC, Overvad K, Jenab M, Fedirko V, Boutron-Ruault MC, Clavel-Chapelon F, Racine A, Kaaks R, Boeing H, Foerster J, Trichopoulou A, Lagiou P, Trichopoulos D, Sacerdote C, Sieri S, Palli D, Tumino R, Panico S, Siersema PD, Peeters PH, Lund E, Barricarte A, Huerta JM, Molina-Montes E, Dorronsoro M, Quiros JR, Duell EJ, Ye W, Sund M, Lindkvist B, Johansen D, Khaw KT, Wareham N, Travis RC, Vineis P, Bueno-de-Mesquita HB, Riboli E. Plasma antibodies to oral bacteria and risk of pancreatic cancer in a large European prospective cohort study. Gut. 2013 Dec;62(12):1764-70. doi: 10.1136/gutjnl-2012-303006. Epub 2012 Sep 18. PMID 22990306
- [Result] Vogtmann E, Han Y, Caporaso JG, Bokulich N, Mohamadkhani A, Moayyedkazemi A, Hua X, Kamangar F, Wan Y, Suman S, Zhu B, Hutchinson A, Dagnall C, Jones K, Hicks B, Shi J, Malekzadeh R, Abnet CC, Pourshams A. Oral microbial community composition is associated with pancreatic cancer: A case-control study in Iran. Cancer Med. 2020 Jan;9(2):797-806. doi: 10.1002/cam4.2660. Epub 2019 Nov 21. PMID 31750624